CLINICAL TRIAL: NCT04103372
Title: Pre-therapeutic MRI Assessment of Early-Stage Rectal Cancer and Significant Rectal Polyps to Avoid Major Resectional Surgery
Acronym: PRESERVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Pelican Cancer Foundation (Other); RM Partners West London Cancer Alliance (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: DOCUMAS 24HH8769
Record Dates: First submitted 2019-09-05; First posted 2019-09-25 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Rectal Cancer; Colo-rectal Cancer
Keywords: early stage; early phase; Endoscopic Mucosal Resection; Endoscopic Submucosal Dissection; Histopathological Staging; MDT Decision Making; MRI Staging; Quality of Life; Radiotherapy; Rectal preservation; Shared decision making; Significant Rectal Polyps; Transanal Endoscopic Microsurgery; Transanal Minimally Invasive Surgery
MeSH Terms: conditions — Rectal Neoplasms; Colonic Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: Multicentre, stepped-wedge cluster randomised trial. This pilot study will run for 9 months and utilise a stepped wedge cluster randomised controlled trial design (including transition period). Sites will enter data from the diagnostic and treatment pathways of all rectal cancer patients who are eligible for primary surgical treatment, eg those radiologically staged as less than or equal to T3b or with confirmed as less than or equal to pT2N0 pathological staging.
  Prior to the trial opening the participating sites will be randomly allocated a number, which will determine the number of months the site will remain in the control and then subsequently the intervention phase of the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm Schedule (No Intervention): All sites will begin in the Control arm, with patients recruited to the Control Arm Schedule. Clinical investigations prior to treatment, during treatment, after surgery and during further treatment should be performed as per standard clinical practice and as clinically indicated. Each site will transition to the Intervention arm at a month prescribed by their randomised cluster, and from that point patients are recruited to the Intervention Arm Schedule . Patients will be recruited to either the Control or Intervention arms dependent on which arm is in progress at the site at the time of recruitment. There will be no crossover of patients between the arms at any point.
- Intervention Arm Schedule (Experimental): Each site will transition to the Intervention arm at a month prescribed by their randomised cluster, and from that point patients are recruited to the Intervention Arm Schedule . The transition period lasts one month during which recruitment is halted and two interventions implemented:
  1. MRI scans will be recommended for all rectal polyps ≥20mm in size, or with other features suspicious of malignancy, prior to removal. This is designed to reduce the numbers of Early Rectal Cancers missed in endoscopy.
  2. Radiologist training in the use of the PRESERVE mrSRT for suspected Early Rectal Cancer.
  Patients will be recruited to either the Control or Intervention arms dependent on which arm is in progress at the site at the time of recruitment. There will be no crossover of patients between the arms at any point.
  Interventions: Diagnostic Test: MRI scan; Other: Radiologist training

INTERVENTIONS:
Diagnostic Test: MRI scan — MRI scans will be recommended for all rectal polyps ≥20mm in size, or with other features suspicious of malignancy, prior to removal. This is designed to reduce the numbers of Early Rectal Cancers missed in endoscopy.
  Arms: Intervention Arm Schedule
Other: Radiologist training — Radiologist training in the use of the PRESERVE mrSRT for suspected Early Rectal Cancer.
  Arms: Intervention Arm Schedule

SUMMARY:
When a patient is diagnosed with a rectal (bowel) polyp or cancer, radiology doctors read MRI scans to describe how deeply the cancer invades into the bowel wall (this is the 'stage' of the cancer). In this project, we will teach radiologists to find more early-stage rectal cancers. These are cancers that have only grown partially into the bowel wall. If we succeed, more patients could have these lesions removed by a local procedure that preserves the bowel and avoids the risks and complications of major surgery.

We have developed a new method for radiology doctors to read MRI scans, which is more accurate than current practice. Currently only 3/10 of early rectal cancers are found by radiologists but by using our MRI reading system, 9/10 patients can be accurately identified as having early rectal cancer. We have proven that we can teach this method to other radiology doctors whose reports help to accurately inform patients of all possible treatment options, so they can be offered the option of a local procedure.

In this initial work we will train radiology doctors in our MRI reading method in 20 hospitals. We will compare MRI reports before and after training to see if an accurate reading method improves treatments choices for patients. We will also determine whether more patients have local procedures after our training. The results of this initial work will help us to apply for national funding for a trial that we can quickly roll out to all NHS hospitals.

DETAILED DESCRIPTION:
Many patients diagnosed with Early Rectal Cancer (ERC) are currently over-treated. Most patients with confirmed ERC will undergo an MRI, but some are not correctly identified in endoscopy and immediately removed. Of those who undergo MRI, 69% are over-staged and undergo major surgery or unnecessary radiotherapy when local excision surgery to preserve the patients rectum, and quality of life, would have been possible. <10% of patients with ERC are staged accurately and offered local excision, with the majority who are staged as ERC on MRI still undergoing major surgery, likely due to uncertainty in the staging report.

Prof Gina Brown developed a more accurate radiological staging system (PRESERVE) or ERC, whereby T2 tumours are identified and classified according to the degree of preservation of the individual layers of the rectal wall. It has been shown that PRESERVE enabled better identification of ERC suitable for local excision from the expected 30% to 89% accuracy. This improved accuracy was replicated in a further study by training a cohort of 12 radiologists. It is predicted that wider adoption of PRESERVE will result in increased organ-preserving surgery from the current rates of 10% to >50%.

ELIGIBILITY:
Inclusion Criteria:

1. Have a rectal tumour or suspected tumour less than or equal to T3b on MRI stage or pT2 or less after excision, or 20mm or more on endoscopy with suspicion of malignancy
2. Be aged 16 years or over

Exclusion Criteria:

1. Have metastatic disease at time of initial staging
2. Have a biopsy-proven rectal malignancy which is not adenocarcinoma
3. Are contraindicated for MRI

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Impact of a training intervention on the accuracy of the tumour staging diagnosis through systematic reporting approach to MRI scans against current (pre intervention) practice. | 1 year
  Comparison of the proportion of patients with early rectal cancer who are diagnosed by pathology vs those staged as such by MRI, before and after the intervention.

SECONDARY OUTCOMES:
Proportion of patients with technically adequacate scans before and after intervention | 1 year
  Proportion of patients scanned with high resolution MR in the correct planes
Proportion of primary tumour characterised by morphology and other features associated with malignancy before and after intervention | 1 year
  Proportion of reports where primary tumour has been characterised by morphology before and after intervention in i) endoscopy, ii) radiology reports before and after intervention
Proportion of MRI reports with T substage given before and after intervention | 1 year
  Proportion of reports where T substage of primary tumour has been recorded before and after intervention
Number of patients identified on imaging as suitable for rectal preservation by local excision | 1 year
  Proportion of imaging reports where suitable patients are identified on the report as suitable for rectal preservation by local excision being identified by the radiologist on the report before and after intervention
Number of patients identified by MDT as suitable for rectal preservation by local excision | 1 year
  Proportion of MDT decisions where patients suitable for rectal preservation by local excision are identified and comparison of treatments offered to patients by the MDT, before and after the intervention
Correlation of accuracy in the identification of safe plane of excision for rectal preservation by the radiologist | 1 year
  Proportion of patients with >1mm muscularis preserved on histopathology identified as such by the radiologist before and after intervention Proportion of patients with >1mm submucosa preserved on histopathology identified as such by the radiologist before and after intervention Proportion of patients undergoing TME that have <1mm muscularis preserved on histopathology identified as such by the radiologist before and after intervention
Numebr of patients with R0 by local excision or TME as appropriate | 1 year
  Proportion of patients with R0 that have >1mm muscularis preserved on histopathology identified as such by the radiologist before and after intervention Proportion of patients with R0 that have>1mm submucosa preserved on histopathology identified as such by the radiologist before and after intervention Proportion of patients undergoing TME with R0 that have <1mm muscularis preserved on histopathology identified as such by the radiologist before and after intervention
Qualitative EORTC QLQ-CR29 Questionnaire on Quality of Life of patients undergoing local excision vs major surgery | 1 year, 3 years, 5 years
  Comparison of QoL EORTC QLQ-CR29 scores before and after intervention. Questions relate to difficulty in performing every day tasks answers are rated 'Not at all' 'A Little' 'Quite a Bit' 'Very Much'
Qualitative EORTC QLQ-CR30 Questionnaire on Quality of Life of patients undergoing local excision vs major surgery | 1 year, 3 years, 5 years
  Comparison of QoL EORTC QLQ-CR30 scores before and after intervention. Questions relate to the presences of symptoms over the previous week answers are rated 'Not at all' 'A Little' 'Quite a Bit' 'Very Much'
Qualitative LARS Questionnaire on Quality of Life of patients undergoing local excision vs major surgery | 1 year, 3 years, 5 years
  Comparison of LARS scores before and after intervention. Questions relate to bowel function answers are rated 'Not at all' 'A Little' 'Quite a Bit' 'Very Much'
Qualitative Questionnaire on Quality of Life of patients undergoing local excision vs major surgery | 1 year, 3 years, 5 years
  Comparison of self evaluation of overall health and quality of life scores before and after intervention. Answers are rated from 1 very poor to 7 excellent
Comparison of total costs of procedures performed between patients undergoing local excision surgery to those undergoing major surgery | 1 year
  Comparison of total costs of hospital procedures performed based on individual pathways before and after intervention
Comparison of inpatient costs between patients undergoing local excision surgery to those undergoing major surgery | 1 year
  Comparison of cost of inpatient episodes based on individual pathways before and after intervention
Comparison of total cost of outpatient visits between patients undergoing local excision surgery to those undergoing major surgery | 1 year
  Comparison of total cost of outpatient episodes based on individual pathways before and after intervention
Comparison of total community costs between patients undergoing local excision surgery to those undergoing major surgery | 1 year
  Comparison of total cost of treatments delivered in the community based on individual pathways before and after intervention
Number of patients without disease and/or without stoma between patients undergoing local excision surgery, compared to those undergoing major surgery | 1 year, 3 years, 5 years
  DFS and stoma free survival in patients based on individual pathways before and after intervention
Assessment results for the effectiveness of mrSRT after a year from training | 1 year
  Determine longevity of training by assessment of radiologists trained with the PRESERVE mrSRT accuracy 1 year after training
Identification of histopathological biomarkers to improve selection of patients who can undergo rectal preserving strategies for Early Recal Cancer | 2 months, 1 year, 3 years, 5 years
  Comparison of relative % histopathological biomarkers screening panels between patients identified on imaging as suitable for rectal preservation by local excision being identified by the radiologist on the report before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Gina Brown, MD, Principal Investigator — Imperial College London
Locations (23):
- United Kingdom (23):
  - Royal Berkshire Hospital, Reading, Berkshire
  - Buckinghamshire Healthcare Nhs Trust, Amersham, Buckinghamshire
  - University College London Hospitals Nhs Foundation Trust, London, Greater London
  - King'S College Hospital Nhs Foundation Trust, London, Greater London
  - West Middlesex Hospital, London, Greater London
  - Imperial College Healthcare Nhs Trus, London, Greater London
  - The Hillingdon Hospitals Nhs Foundation Trust, Uxbridge, Greater London
  - Hampshire Hospitals Nhs Foundation Trust, Basingstoke, Hampshire
  - Southampton General Hospital, Southampton, Hampshire
  - Kent & Canterbury Hospital, Canterbury, KENT
  - Maidstone Hospital, Maidstone, KENT
  - Westmorland General Hospital, Kendal, Lancashire
  - Leicester Royal Infirmary, Leicester, Leicestershire
  - St George'S Hospital, Tooting, London
  - John Radcliffe Hospital, Oxford, Oxfordshire
  - Nhs Staffordshire and Stoke-on-Trent Integrated Care Board, Stafford, Staffordshire
  - Frimley Health Nhs Foundation Trust, Camberley, Surrey
  - St Helier Hospital, Carshalton, Surrey
  - Kingston Hospital Nhs Foundation Trust, Kingston upon Thames, Surrey
  - Croydon Health Services Nhs Trust, Thornton Heath, Surrey
  - Tonna Hospital, Swansea, Wales
  - Salisbury District Hospital, Salisbury, Wiltshire
  - St Marks Bowel Cancer Screening Centre, Harrow

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Detering R, van Oostendorp SE, Meyer VM, van Dieren S, Bos ACRK, Dekker JWT, Reerink O, van Waesberghe JHTM, Marijnen CAM, Moons LMG, Beets-Tan RGH, Hompes R, van Westreenen HL, Tanis PJ, Tuynman JB; Dutch ColoRectal Audit Group*. MRI cT1-2 rectal cancer staging accuracy: a population-based study. Br J Surg. 2020 Sep;107(10):1372-1382. doi: 10.1002/bjs.11590. Epub 2020 Apr 16. PMID 32297326
- [Background] Balyasnikova S, Read J, Wotherspoon A, Rasheed S, Tekkis P, Tait D, Cunningham D, Brown G. Diagnostic accuracy of high-resolution MRI as a method to predict potentially safe endoscopic and surgical planes in patients with early rectal cancer. BMJ Open Gastroenterol. 2017 Aug 14;4(1):e000151. doi: 10.1136/bmjgast-2017-000151. eCollection 2017. PMID 29259791
- See also: National Bowel Cancer Audit. Annual Report 2022 [Internet]. Leeds: NBOCA; 2022 — https://www.nboca.org.uk/content/uploads/2023/01/NBOCA-2022-Final.pdf